CLINICAL TRIAL: NCT02651623
Title: A Phase 1, Single Center Randomized, Three-way Crossover, Double-blinded, Placebo- And Moxifloxacin-controlled Thorough Qt (Tqt) Study To Determine The Effects Of Sertraline (Zoloft (Registered)) On The Cardiac Repolarization In Healthy Subjects
Brief Title: Study to Evaluate The Effect Of Sertraline on the Cardiac Repolarization in Healthy Subjects
Acronym: Zoloft
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: A0501104; 2015-000103-47 (EudraCT Number); TQT (Other: Alias Study Number)
Record Dates: First submitted 2015-11-20; First posted 2016-01-11 (Estimated); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Healthy
MeSH Terms: interventions — Sertraline; Bulk Drugs; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Sertraline (Experimental): Maximum dose of 400 mg/day (200 mg BID given at approximately 12 hours apart) sertraline, dose titrated from a starting single dose (QD) of 50 mg in the morning on Day 1 followed by BID doses administered on Days 2 through 14 (Day 14 morning dose only) will be administered
  Interventions: Drug: Sertraline
- Moxifloxacin (Active Comparator): 400 mg single dose of moxifloxacin (Avelox®) administered on Day 14
  Interventions: Drug: Moxifloxacin
- Drug - Placebo (Placebo Comparator): placebo - placebo administered on Days 1 through 14
  Interventions: Drug: Drug - Placebo

INTERVENTIONS:
Drug: Sertraline — Multiple doses of sertraline for 14 days
  Other Names: active drug
  Arms: Sertraline
Drug: Moxifloxacin — A single dose of 400 mg Moxifloxacin
  Other Names: Positive control
  Arms: Moxifloxacin
Drug: Drug - Placebo — Placebo administered for 14 days
  Other Names: Placebo control
  Arms: Drug - Placebo

SUMMARY:
The purpose of this study is to demonstrate a lack of effect of sertraline on QTc intervals relative to time-matched placebo in healthy subjects

DETAILED DESCRIPTION:
Evaluate multiple doses of 400 mg per day of sertraline on QTc, and evaluate the safety and tolerability of sertraline in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lbs).

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing).

Risk factors for QT prolongation or torsades de pointes

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2016-01; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Postdose QTcF (Fridericia's correction) intervals | 0 to 72 hours

SECONDARY OUTCOMES:
Averse events, vital signs, physical examinations and abnormal laboratory for safety assessments (safety and tolerability) | Through study completion, an average of 3 months
Relationship between QTc prolongation and measured sertraline/metabolite plasma concentrations | 0 to 72 hours

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Clinical Research Unit, Brussels, Belgium

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0501104&StudyName=A+Phase+1%2C+Single+Center+Randomized%2C+Three-way+Crossover%2C+Double-blinded%2C+Placebo-+And+Moxifloxacin-controlled+Thorough+Qt+%28tqt%29+Study+To+Determine+The+Effects+Of+Sertraline+%28zoloft+%28registered%29%29+On+The+Cardiac+Repolarization+In+Healthy+Subjects